CLINICAL TRIAL: NCT02757742
Title: A Quantitive Late Gadolinium Enhancement(LGE) Mass Based Tool for Risk Prediction of Sudden Cardiac Death(SCD) in Non-ischemic Cardiomyopathy(NICM) Patients With Severe Cardiac Dysfunction
Brief Title: Quantitive LGE Mass in Prediction of SCD in NICM Patients With Severe Cardiac Dysfunction
Status: Completed | Type: Observational
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Fan Xiaohan, Associated director, head of Cardiology,Principal Investigation, Clinical Professor, Fu Wai Hospital, Beijing, China
Other Study IDs: NICM-002-FW
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Cardiomyopathy
Keywords: sudden cardiac death; ventricular arrhythmias; cardiopathy; late gadolinium enhancement
MeSH Terms: conditions — Cardiomyopathies; Death, Sudden, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-ischemic cardiomyopathy: Non-ischemic cardiomyopathy patients with baseline cardiac magnetic resonance LVEF≤35%

SUMMARY:
The purpose of this study is to establish a quantitative LGE mass based scoring system (including LGE mass on cardiac magnetic resonance , clinical features, specific medical histories, et al) for risk prediction of sudden cardiac death in non-ischemic dilated cardiomyopathy patients with reduced left ventricular ejection fraction

DETAILED DESCRIPTION:
This is a Single-centered, Prospective, Observational Study. The study design included two phases. In Phase I, the investigators enrolled a set of consecutive patients with non-ischemic cardiomyopathy who performed contrast-enhanced cardiac magnetic resonance at baseline and had severe cardiac dysfunction (defined as cardiac magnetic resonance LVEF equal or less than 35% ) in FuWai Hospital from 2010 to 2013. The investigators collect patients' clinical baseline data and cardiac magnetic resonance specific data(Late gadolinium enhancement mass). All patients were followed up every six month by phone or clinical visits. The primary endpoint was composite of sudden cardiac death(SCD), ventricular arrhythmias(VAs) and SCD/VAs related Implantable Cardioverter defibrillator or cardiac resynchronization therapy-cardioverter defibrillator(ICD/CRTD) shock. The investigators plan to establish a quantitative LGE mass based model (including LGE mass on cardiac magnetic resonance, clinical features, specific medical histories, et al) for risk prediction of sudden cardiac death by analysing the phase I data(1-year model and 3-year model). In Phase II,the investigators will enroll another group of non-ischemic cardiomyopathy(NICM) patients from 2014 to 2015 to testify the risk prediction model(1-year model) the investigators have constructed in phase I. The investigators aim to find the real high risk NICM patients that may suffer from SCD or VAs in those with severe cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Non-ischemic cardiomyopathy patients receiving optimal medical treatment for 3 months; Age range from 10 years to 65 years old； Baseline cardiac magnetic resonance LVEF≤35%

Exclusion Criteria:

* Known associated obstructive coronary Heart disease（including history of myocardial infarction or acute coronary event）； valvular heart disease； malignant carcinoma ； hypertensive heart disease； severe liver or kidney dysfunction ； plan to receiving heart transplantation ； patients refuse to or cannot receive cardiac magnetic resonance ； patients refuse to be followed up ；

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients with non-ischemic cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2010-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Sudden cardiac death(SCD) | Six years
  SCD was defined as cardiac death occured in a short time period (2 hour of symptom), which were assessed by two separated doctors from the central laboratory.
Aborted cardiac arrest | Six years
  Aborted cardiac arrest were defined as patients with ventricular tachycardia, ventricular fibrillation or sudden cardiac death were saved by cardio-pulmonary resuscitation and electric defibrillation.
Documented appropriate ICD therapy for ventricular tachycardia | Six years
  Participants with ICD or CRTD implanted came to the clinic every 6 months for device's programming control. Shock related events were analyzed by two separated experienced electrophysiology doctor(more than 5 years),to identify if the shock is delivered by sustained ventricular tachycardia, ventricular fibrillation and sudden cardiac death.
Documented appropriate ICD therapy for ventricular fibrillation | Six years
  Participants with ICD or CRTD implanted came to the clinic every 6 months for device's programming control. Shock related events were analyzed by two separated experienced electrophysiology doctor(more than 5 years),to identify if the shock is delivered by sustained ventricular tachycardia, ventricular fibrillation and sudden cardiac death.

SECONDARY OUTCOMES:
All-cause death(including cardiac death and non-cardiac death) | six years
  Participants were followed up every 6 months and the survival status of participants were documented(death or not, if the patient was dead, time of death and cause of death were documented)
Heart transplantation | six years
  Participants were followed up every 6 months, if the patients received heart transplantation, the follow ups were terminated and time for heart transplantation were documented.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan Fan, MD,PHD, Principal Investigator — Fu Wai Hospital
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Chan RH, Maron BJ, Olivotto I, Pencina MJ, Assenza GE, Haas T, Lesser JR, Gruner C, Crean AM, Rakowski H, Udelson JE, Rowin E, Lombardi M, Cecchi F, Tomberli B, Spirito P, Formisano F, Biagini E, Rapezzi C, De Cecco CN, Autore C, Cook EF, Hong SN, Gibson CM, Manning WJ, Appelbaum E, Maron MS. Prognostic value of quantitative contrast-enhanced cardiovascular magnetic resonance for the evaluation of sudden death risk in patients with hypertrophic cardiomyopathy. Circulation. 2014 Aug 5;130(6):484-95. doi: 10.1161/CIRCULATIONAHA.113.007094. PMID 25092278
- [Background] Dou K, Zhang D, Xu B, Yang Y, Yin D, Qiao S, Wu Y, Yan H, You S, Wang Y, Wu Z, Gao R, Kirtane AJ. An angiographic tool for risk prediction of side branch occlusion in coronary bifurcation intervention: the RESOLVE score system (Risk prEdiction of Side branch OccLusion in coronary bifurcation interVEntion). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):39-46. doi: 10.1016/j.jcin.2014.08.011. PMID 25616815
- [Background] Zhang S, Singh B, Rodriguez DA, Chasnoits AR, Hussin A, Ching CK, Huang D, Liu YB, Cerkvenik J, Willey S, Kim YH. Improve the prevention of sudden cardiac arrest in emerging countries: the Improve SCA clinical study design. Europace. 2015 Nov;17(11):1720-6. doi: 10.1093/europace/euv103. Epub 2015 Jun 1. PMID 26037794
- [Background] Zhang S. Sudden cardiac death in China: current status and future perspectives. Europace. 2015 Oct;17 Suppl 2:ii14-8. doi: 10.1093/europace/euv143. PMID 26842111
- [Background] Tateishi E, Noguchi T, Goto Y, Morita Y, Ishibashi-Ueda H, Yamada N, Kanzaki H, Nishimura K, Miyamoto Y, Anzai T, Ogawa H, Yasuda S. Prognostic impact of blood pressure response plus gadolinium enhancement in dilated cardiomyopathy. Heart. 2015 May 15;101(10):774-80. doi: 10.1136/heartjnl-2014-307007. Epub 2015 Mar 11. PMID 25761994
- [Background] Duan X, Li J, Zhang Q, Zeng Z, Luo Y, Jiang J, Chen Y. Prognostic value of late gadolinium enhancement in dilated cardiomyopathy patients: a meta-analysis. Clin Radiol. 2015 Sep;70(9):999-1008. doi: 10.1016/j.crad.2015.05.007. Epub 2015 Jun 23. PMID 26116301
- [Background] Kang Y, Cheng L, Cui J, Li L, Qin S, Su Y, Mao J, Gong X, Chen H, Pan C, Shen X, He B, Shu X. A new score system for predicting response to cardiac resynchronization therapy. Cardiol J. 2015;22(2):179-87. doi: 10.5603/CJ.a2014.0089. Epub 2014 Nov 27. PMID 25428735
- [Background] Sakamoto N, Sato N, Talib AK, Sugiyama E, Minoshima A, Tanabe Y, Fujino T, Takeuchi T, Akasaka K, Saijo Y, Kawamura Y, Hasebe N. Late Gadolinium Enhancement on Cardiac MRI Correlates with QT Dynamicity Represented by QT/RR Relationship in Patients with Ventricular Arrhythmias. Ann Noninvasive Electrocardiol. 2016 Mar;21(2):126-35. doi: 10.1111/anec.12280. Epub 2015 Jun 24. PMID 26104916